CLINICAL TRIAL: NCT01743300
Title: The Influence of Genotype/Phenotype, Grapefruit Juice and Orange Juice on the Pharmacokinetics of Sunitinib (Sutent, SU011248) in Patient With Imatinib Resistant Gastrointestinal Stromal Cell Tumor (GIST) or Metastatic Renal Cell Carcinoma
Brief Title: The Influence of Phenotype, Grapefruit Juice and Orange Juice on the Pharmacokinetics of Sunitinib in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Hans Gelderblom, Prof., Leiden University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: P07.111
Record Dates: First submitted 2012-11-15; First posted 2012-12-06 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: sunitinib; pharmacokinetics; phenotyping; interaction
MeSH Terms: interventions — Sunitinib; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Grapefruit juice arm (Active Comparator): The grapefruit juice will be administered 3 times per day for 1 period of 3 days in the 4th week of treatment
  Interventions: Drug: Sunitinib; Drug: Midazolam; Other: Grapefruit juice
- Orange juice (Active Comparator): The orange juice will be administered 3 times per day for 1 period of 3 days in the 4th week of treatment.
  Interventions: Drug: Sunitinib; Drug: Midazolam; Other: Orange juice

INTERVENTIONS:
Drug: Sunitinib — All patients receive once daily 50 mg sunitinib for 6 weeks in the registered schedule of 4 weeks on two weeks off treatment.
  Other Names: sutent
Drug: Midazolam — All patients receive three times midazolam 7,5 mg on PK day 1,2, and 3 e.g. between day 14-21 of treatment, on day 28 of treatment and on day 42 of treatment.
  Other Names: Dormicum
Other: Orange juice — The orange juice will be administered 3 times per day for 1 period of 3 days in the 4th week of treatment with sunitinib, just before PK day 2 on day 28 of treatment
  Arms: Orange juice
Other: Grapefruit juice — The grapefruit juice will be administered 3 times per day for 1 period of 3 days in the 4th week of treatment with sunitinib, just before PK day 2 on day 28 of treatment
  Arms: Grapefruit juice arm

SUMMARY:
In this prospective pharmacokinetic we investigate the following topics:

* The influence of grapefruit juice and orange juice on the steady-state pharmacokinetics of sunitinib in cancer patients
* The influence of sunitinib on the pharmacokinetics of midazolam in cancer patients
* The relationship between Cytochrome-P450-3A4 (CYP3A4) phenotype, as assessed using the midazolam clearance test, and the steady-state pharmacokinetics of sunitinib in cancer patients
* The effect of grapefruit juice and orange juice on CYP3A4 metabolism

DETAILED DESCRIPTION:
This is a prospective pharmacokinetic study in two groups of 10 adult patients with imatinib-resistant gastro-intestinal stromal cell tumor or metastatic renal cell carcinoma treated with sunitinib for at least one month.

Patients are treated at the recommended United States Food and Drug Administration approved schedule of oral sunitinib administered at 25-50 mg per day for 4 weeks, in cycles of six weeks. Four weeks of treatment with sunitinib, 25-50 mg per day followed by a 2 weeks off period. In the absence of disease progression, administration of sunitinib will continue.

Within one month of the start of the study, patients will be requested to refrain from drinking grapefruit and orange juice. The study will take place in 1 sunitinib treatment cycle of 6 weeks (4 weeks of treatment with sunitinib (week 1-4) and 2 weeks off period (week 5 and 6). The grapefruit juice or orange juice will be administered 3 times per day for 1 period of 3 days in the 4th week of treatment with sunitinib.

The first sunitinib (total drug) pharmacokinetics day will be performed after steady-state sunitinib levels are reached, meaning at least 14 days after starting sunitinib 25 - 50 mg per day treatment (week 3 in the treatment cycle of sunitinib). On this first pharmacokinetic day a dose of midazolam 7.5 mg will be given at the same time as the sunitinib dose, to observe the effect of sunitinib on CYP3A4 capacity. Before the second pharmacokinetic day (day 28 of sunitinib treatment) the patient will drink 3 times a day a glass of grapefruit juice or orange juice for three consecutive day.Patients will be assigned either to a grapefruit juice or orange juice arm. On this second pharmacokinetic day the patient again will use a dose of midazolam at the sam time as the sunitinib dose, to observe the effect of grapefruit juice or orange juice on the metabolic capacity pf CYP3A4. The third pharmacokinetic day will take place at the end of week 6 of the treatment cycle, the second week of the 2 week off period. The patient will receive a single oral dose of midazolam 7.5mg, followed by midazolam pharmacokinetics to determine the base-line CYP3A phenotypic expression. Pharmacokinetic parameters based on measurement in plasma samples will be compared between the treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with imatinib-resistant gastro-intestinal stromal cell tumor or metastatic renal cell carcinoma treated with sunitinib at a dose level of 25-50 mg sunitinib per day in a 4 weeks on/2 weeks off schedule.
* Age at least 18 years
* WHO performance status < 2.
* At least 4 weeks since last chemotherapy, hormonal, or radiation therapy.
* A life expectancy of at least 12 weeks.
* Patients must have an adequate functional reserve as defined by: hemoglobin > 6.0 mmol/L, White Blood Count > 3.0 x 109/L, neutrophils > 1.5 x 109/L, platelets > 100 x 109/L, creatinine clearance > 60 mL/min, bilirubin within normal limits, Alanine transaminase and aspartate transaminase < 2.5 times the upper limit of normal (unless due to liver metastases, then < 5 times the upper limit of normal.
* Written informed consent.

Exclusion Criteria:

* Patients with hematological malignancies
* Concurrent other chemotherapy, immunotherapy, or radiotherapy.
* Concurrent use of other substances known or likely to interfere with the pharmacokinetics of sunitinib (e.g., ketoconazole, cyclosporine A).
* Use of drugs, herbal preparations and/or dietary supplements known to influence the expression of CYP3A (e.g., phenytoin, rifampicin, St. John's wort, garlic supplements, milk thistle) within the preceding 2 weeks.
* Present clinical signs of symptoms of brain and/or leptomeningeal metastases confirmed by CT or MRI brain scan. A patient with brain and/or leptomeningeal metastases may be included only if he/she is asymptomatic on neurological examination and is not receiving corticosteroid therapy to control symptoms.
* Patients with uncontrolled infection.
* Concurrent severe medical problems unrelated to the malignancy that would limit full compliance with the study or expose the patient to extreme risk.
* Patients with pre-existing cardiac disease, including clinical congestive heart failure, cardiac arrhythmias requiring treatment, or a myocardial infarction within the preceding 3 months.
* Patients who have received another investigational drug within 30 days or 5 half-lives prior to entry in the study (whichever is longer).
* History of allergic reaction to compounds chemically related to sunitinib.
* Patients who are pregnant or breastfeeding.
* Patients of childbearing potential, not practicing adequate contraception.
* Patients that are unable to ingest oral medication and/or are known with gastric emptying disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The influence of grapefruit juice and orange juice on the steady state area under the curve (AUC) of sunitinib in cancer patients | Patients will be included for 42 days into the study. Within these 42 days, 3 PK measuring days are planned (see also description)
  Subjects will receive sunitinib in the registered schedule of 4 weeks "on" (28 days) 2 weeks "off" (14 days).Sunitinib steady state is reached after 14 days. Additionally patients receive grapefruit juice on day 25-27 of treatment. To determine the influence of grapefruit juice, sunitinib pharmacokinetics (PK) will be assessed on PK day 1, which will be between treatment day 14-20 (without grapefruit juice) and on PK day 2 on day 28 of treatment (after taking grapefruit juice for 3 days).
The feasibility of midazolam as a phenotyping probe for sunitinib exposure (area under concentration time curve)in cancer patients | Patients will be included for 42 days into the study. Within these 42 days, 3 PK measuring days are planned (see also description)
  Subjects will receive sunitinib in the registered schedule of 4 weeks "on" (28 days) 2 weeks "off" (14 days).Sunitinib steady state is reached after 14 days. To determine the feasibility of midazolam as a phenotyping probe, sunitinib PK from PK day 1, which is between treatment day 14-20 and the PK of midazolam from PK day 3 on day 42 of treatment (the end of the wash out period of sunitinib) will be determined.

SECONDARY OUTCOMES:
The effect of grapefruit juice and orange juice on CYP3A4 metabolism | Patients will be included for 42 days into the study. Within these 42 days, 3 PK measuring days are planned (see also description)
  Subjects will receive sunitinib in the registered schedule of 4 weeks "on" (28 days) 2 weeks "off" (14 days).Sunitinib steady state is reached after 14 days. Additionally patients receive grapefruit juice on day 25-27 of treatment and midazolam on PK days. To determine the influence of grapefruit juice on CYP 3A4 metabolism, midazolam PK will be assessed on PK day 1, which will be between treatment day 14-20 (without grapefruit juice) and on PK day 2 on day 28 of treatment (after taking grapefruit juice for 3 days).
The influence of sunitinib on CYP3A4 activity | Patients will be included for 42 days into the study. Within these 42 days, 3 PK measuring days are planned (see also description)
  Subjects will receive sunitinib in the registered schedule of 4 weeks "on" (28 days) 2 weeks "off" (14 days).Sunitinib steady state is reached after 14 days. Additionally, patients receive midazolam on PK day 1 (between treatment day 14-20)and PK day 3 (day 42 of treatment,the end of the wash out period of sunitinib). To determine the influence of sunitinib on CYP3A4 activity, midazolam PK of PK day 1 (sunitinib AND midazolam) will be compared to midazolam PK of PK day 3 (midazolam alone)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gelderblom, Principal Investigator — LUMC